CLINICAL TRIAL: NCT05645172
Title: Retention Rate of Acalabrutinib in a Non-interventional Setting
Acronym: RETAIN
Status: Active, not recruiting | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8224R00001
Record Dates: First submitted 2022-11-10; First posted 2022-12-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Chronic Lymphocytic Leukaemia (CLL)
Keywords: Acalabrutinib
MeSH Terms: conditions — Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: adult CLL patients (≥ 18 years of age) newly prescribed with acalabrutinib according to clinical routine will be included independent of the patient age, disease stage, existence of genetic risk factors, comorbidities, therapy line, and of the application as combination therapy with obinutuzumab or as monotherapy.

SUMMARY:
Retention rate of acalabrutinib in a non-interventional setting. This is a prospective, multicentre, non-interventional study to collect real-world data on retention rates of CLL patients prescribed with acalabrutinib in Germany.

DETAILED DESCRIPTION:
This observational study will prospectively assess acalabrutinib therapy retention of CLL patients one year and 2 years after treatment initiation with acalabrutinib in routine clinical practice. Furthermore, therapy adherence, treatment efficacy, overall survival, and QoL to analyse the possible influence of psychological aspects of the patient-based disease perception, a four-group-segmentation for acceptance and perceived control of the health state will be conducted. Finally, disease-, treatment-, and patient-specific factors possibly affecting therapy retention will be analysed: sociodemographic factors, disease and treatment characteristics, comorbidities, therapy adherence, treatment effectiveness, safety, QoL, and psychological segmentation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of CLL
* Ability to understand the study concept and to regularly complete patient questionnaires from physical, mental, and linguistic perspectives
* Decision to start therapy with acalabrutinib according to the current SmPC. For previously untreated patients as continuous therapy with or without obinutuzumab. OR For patients with at least one prior CLL therapy as continuous monotherapy.
* Provision of signed informed consent form

Exclusion Criteria:

* Current or planned participation in an interventional clinical trial
* Contraindications to treatment with acalabrutinib according to the current SmPC
* Pregnancy or breast feeding
* Disease progression on prior BTKi therapy
* Start of acalabrutinib therapy more than 28 days prior to enrolment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CLL patients with a newly initiated acalabrutinib treatment in routine clinical practice are planned to be included from approximately 75 sites in Germany over a recruitment period of 16 months.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2022-12-12 (Actual); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-15 (Estimated)

PRIMARY OUTCOMES:
Retention rate of CLL | 1 year
  The primary outcome of this study is the retention rate of CLL patients receiving acalabrutinib in clinical practice after 1 year (= ratio of the number of patients still being prescribed acalabrutinib after 1 year to the number of patients at risk). Cases of death, ongoing treatment interruption, and lost to follow-up will be counted as patients not still being prescribed with acalabrutinib.

SECONDARY OUTCOMES:
Retention rate of CLL | 2 years
  The secondary outcome is the retention rate of CLL patients receiving acalabrutinib in clinical practice after 2 years.
General treatment adherence | assessed at baseline and 6, 12, and 24 months after start of acalabrutinib treatment
  General treatment adherence will be assessed over the whole observational period by the self-reported, 8-item structured MMAS-8 questionnaire.
reasons for and duration of therapy interruptions | time from first prescription until therapy interruptions; assessed up to 40 months
  Based on acalabrutinib treatment details, the reasons for and duration of therapy interruptions will be calculated and analysed.
TTD | time from start of acalabrutinib treatment until the date of final discontinuation or death; assessed up to 40 months.
  Based on acalabrutinib treatment details, the TTD, defined as the time from first prescription until the date of last intake or death, whichever occurs first, will be calculated and the reasons for therapy discontinuation will be analysed.
TTNT | time from start of acalabrutinib treatment until start of a subsequent CLL treatment; assessed up to 40 months.
  Based on acalabrutinib treatment details, the TTNT, defined as the time of first prescription until start date of the next CLL treatment will be calculated and the reasons for switch of treatment will be analysed. Cases of death will be censored and not considered as TTNT-relevant event.
TTNT-D | time from start of acalabrutinib treatment until start of a subsequent CLL treatment or death; assessed up to 40 months
  Based on acalabrutinib treatment details, the TTNT-D, defined as the time of first prescription until start date of the next CLL treatment or death, whichever occurs first, will be calculated.
Treatment efficacy and PFS | time from start of acalabrutinib treatment until disease progression or death by any cause, whichever occurs first; assessed up to 40 months.
  Treatment efficacy will be analysed by means of the overall treatment response (CR, PR, PRL, judged by the treating physician and recommended to be in accordance with the guidelines of the International Workshop on Chronic Lymphocytic Leukemia (iwCLL), modified for persistent lymphocytosis, the time to and duration of response, the percentage of patients without treatment response (SD, PD), as well as the time of PFS, defined as the time of first prescription until progression of the disease or death by any cause, whichever occurs first.
Overall survival | time from start of acalabrutinib treatment until death by any cause; assessed up to 40 months.
  Overall survival will be calculated as the time from first prescription until death by any cause.
Patient- and disease-specific factors possibly affecting the retention rate | up to 40 months
  Patient- and disease-specific factors possibly affecting the retention rate will be analysed for associations with the following variables:
  - Treatment effectiveness (treatment response, PFS)
Healths-related Quality of Life (HRQoL)-QLQ-C30 | Patient questionnaires will becollected at time points synchronised with regular visits during study, assessed up to 40 months
  The QoL, as measured by the self-reported QLQ-C30 questionnaires, will be assessed at baseline and every quarterly regular follow-up visit thereafter until end of observation. The time course of the QoL will be visualised and the mean difference from baseline until 6, 12, and 24 months after start of therapy will be calculated. Clinical significance will be defined as minimal important differences (MIDs) of at least 10 points (in either direction) for total scores or subscales of the QLQ-C30.
Healths-related Quality of Life (HRQoL)-EQ-5D-5L | Patient questionnaires will becollected at time points synchronised with regular visits during study, assessed up to 40 months
  The QoL, as measured by the self-reported EQ-5D-5L questionnaires, will be assessed at baseline and every quarterly regular follow-up visit thereafter until end of observation. The time course of the QoL will be visualised and the mean difference from baseline until 6, 12, and 24 months after start of therapy will be calculated.
Patient- and disease-specific factors possibly affecting the retention rate | up to 40 months
  Patient- and disease-specific factors possibly affecting the retention rate will be analysed for associations with the following variables:
  - Patient- and disease-specific characteristics (sociodemographic data, disease characteristics and severity, comorbidities (CIRS), comedication).
Patient- and disease-specific factors possibly affecting the retention rate | up to 40 months
  Patient- and disease-specific factors possibly affecting the retention rate will be analysed for associations with the following variables:
  - Treatment adherence (MMAS-8).
Patient- and disease-specific factors possibly affecting the retention rate (Psychological patient segmentation) | at Baseline
  Psychological patient segmentation as determinant for the disease acceptance and disease control will be performed during the baseline visit by using a questionnaire published by Bloem et al. in 2020
Patient- and disease-specific factors possibly affecting the retention rate | up to 40 months
  Patient- and disease-specific factors possibly affecting the retention rate will be analysed for associations with the following variables:
  - Safety (rate, severity, and duration of SAEs and ADRs)

CONTACTS AND LOCATIONS:
Locations (54):
- Germany (54):
  - Research Site, D Ren, Germany
  - Research Site, Herrsching am Ammersee, Germany
  - Research Site, L Rrach, Germany
  - Research Site, M Nchen, Germany
  - Research Site, N Rnberg, Germany
  - Research Site, Neustadt Am R Benberge, Germany
  - Research Site, Saarbr Cken, Germany
  - Research Site, Sindelfinden, Germany
  - Research Site, W Rselen, Germany
  - Research Site, Amberg
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Bad Homburg
  - Research Site, Bad Liebenwerda
  - Research Site, Bautzen
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Dachau
  - Research Site, Delitzsch
  - Research Site, Dessau
  - Research Site, Dortmund
  - Research Site, Erfurt
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Garbsen
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heide
  - Research Site, Herten
  - Research Site, Hof
  - Research Site, Kulmbach
  - Research Site, Laatzen
  - Research Site, Landshut
  - Research Site, Lebach
  - Research Site, Leipzig
  - Research Site, Moers
  - Research Site, Naunhof
  - Research Site, Oldenburg
  - Research Site, Paderborn
  - Research Site, Pasing
  - Research Site, Pirna
  - Research Site, Porta Westfalica
  - Research Site, Potsdam
  - Research Site, Remscheid
  - Research Site, Reutlingen
  - Research Site, Riesa
  - Research Site, Saalfeld
  - Research Site, Schkeuditz
  - Research Site, Schorndorf
  - Research Site, Siegburg
  - Research Site, Straubing
  - Research Site, Twistringen
  - Research Site, Weiden
  - Research Site, Zittau

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home